CLINICAL TRIAL: NCT01576146
Title: A Multicenter Open-label Extension Study to Assess the Long-term Safety and Efficacy of KAI-4169 (Also Known as AMG 416) in the Treatment of Chronic Kidney Disease-Mineral and Bone Disorder in Patients With Secondary Hyperparathyroidism
Brief Title: Open-label Study to Assess the Long-term Safety and Efficacy of Etelcalcetide (Also Known as AMG 416 or KAI-4169) in Patients With Secondary Hyperparathyroidism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early to allow subjects to roll over to study NCT02102204.
Sponsor: KAI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAI-4169-005-01; 20120334 (Other: Amgen, Inc)
Record Dates: First submitted 2012-04-05; First posted 2012-04-12 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Clinical Trial, Phase 2; Renal Dialysis; Secondary Hyperparathyroidism; Chronic kidney disease-mineral and bone disorder; Parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etelcalcetide (Experimental): Participants received a bolus IV injection of etelcalcetide 3 times a week (TIW) at the end of each hemodialysis session for up to 144 weeks in the extension study. The starting dose was the same as the final dose administered in the parent study (20120331); the dose was adjusted per protocol-specified guidelines to achieve or maintain parathyroid hormone values in the 150 to 300 pg/mL range.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered as an intravenous bolus three times a week at the end of each hemodialysis session at dosages up to a maximum of 15 mg.
  Other Names: KAI-4169; AMG 416; Parsabiv™

SUMMARY:
The purpose of this study is to evaluate the long term safety and efficacy of thrice weekly intravenous (IV) administration of etelcalcetide in the treatment of secondary hyperparathyroidism (SHPT) in patients receiving hemodialysis who had completed 12 weeks of treatment with etelcalcetide in parent study 20120331 (KAI-4169-005; NCT01414114).

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent.
* Subject completed the 12 week treatment phase in the parent study study 20120331 ( KAI-4169-005; NCT01414114).

Exclusion Criteria:

* Subject pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M D, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label extension study was conducted at 5 centers in the United States. Eligible participants must have completed 12 weeks of treatment in parent study 20120331 (KAI-4169-005; NCT01414114).
Pre-assignment Details: This study consisted of 40 weeks of treatment in extension period 1 followed by 2 years of additional treatment in extension period 2.
  The Sponsor ended the study early. Participants had the opportunity to rollover into another open-label extension study 20130213 (NCT02102204).
Groups:
- Etelcalcetide: Participants received a bolus intravenous (IV) injection of etelcalcetide 3 times a week (TIW) at the end of each hemodialysis session for up to 144 weeks in the extension study. The starting dose was the same as the final dose administered in the parent study (20120331); the dose was adjusted per protocol-specified guidelines to achieve or maintain parathyroid hormone values in the 150 to 300 pg/mL range.
Period: Extension Period 1
Arm/Group | Etelcalcetide
Started | 30
Completed | 20
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Parathyroidectomy | 1
Not completed — Renal Transplant | 1
Period: Extension Period 2
Arm/Group | Etelcalcetide
Started | 17 (Three participants who completed Extension Period 1 did not enroll in Period 2)
Completed | 0
Not Completed | 17
Not completed — Sponsor Decision | 13
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Renal Transplant | 1
Not completed — Treatment Not Resumed Within 8 Weeks | 1

BASELINE CHARACTERISTICS:
Population: Baseline was defined as the baseline of the parent study, 20120331.
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race [Count of Participants; unit: Participants]
  Black (or African American) | 18
  White | 12
Ethnicity [Count of Participants; unit: Participants]
  Hispanic/Latino | 6
  Not Hispanic/Latino | 24
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 862.1 (672.0)
Serum Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] | 10.21 (0.53)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 5.77 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From the first dose of study drug in the parent study (20120331) through 30 days after the last dose in the extension study; actual median duration of treatment was 439 days.
Population: Participants who received at least one dose of etelcalcetide in the extension study
Measure: Number; unit: participants
Groups:
- Etelcalcetide: Participants received a bolus IV injection of etelcalcetide 3 times a week at the end of each hemodialysis session for up to 144 weeks in the extension study. The starting dose was the same as the final dose administered in the parent study (20120331); the dose was adjusted per protocol-specified guidelines to achieve or maintain parathyroid hormone values in the 150 to 300 pg/mL range.
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 30
participants
  Any adverse event (AE) | 30
  Serious adverse events | 18
  Treatment-related adverse events | 13
  Treatment-related serious adverse events | 1
  AEs leading to discontinuation of treatment | 3
  Fatal adverse events | 4

2. Secondary Outcome: Percent Change From Baseline in Parathyroid Hormone
Description: Baseline was defined as the average of 3 predialysis results obtained within 3 weeks before the first dose of etelcalcetide in the parent study (20120331).
  The week numbering for this study continued from the parent study 20120331 hence the first measurement for all parameters in the extension study started at week 13.
Time Frame: Baseline (of the parent study 20120331) and Weeks 13, 26 and 52
Population: The full analysis set (all participants who received at least 1 dose during the extension study) with data collected on or before the last non-missing dose of etelcalcetide (defined as on-treatment approach).
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 30
percent change
  Week 13 | -57.8 (4.0)
  Week 26: number analyzed (Participants) | 26
  Week 26 | -61.0 (5.2)
  Week 52: number analyzed (Participants) | 20
  Week 52 | -51.7 (6.8)

3. Secondary Outcome: Percent Change From Baseline in Serum Corrected Calcium
Description: Baseline was defined as the average of 3 predialysis results obtained within 3 weeks before the first dose of study drug in the parent study (20120331).
  The week numbering for this study continued from the parent study 20120331; the first measurement for all parameters in the extension study started at week 13.
Time Frame: Baseline and Weeks 13, 26 and 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 30
percent change
  Week 13 | -16.16 (1.26)
  Week 26: number analyzed (Participants) | 25
  Week 26 | -13.09 (1.02)
  Week 52: number analyzed (Participants) | 20
  Week 52 | -11.69 (1.38)

4. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus
Description: as for outcome 3
Time Frame: Baseline and Weeks 13, 26 and 52
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 30
percent change
  Week 13 | -10.39 (3.85)
  Week 26: number analyzed (Participants) | 25
  Week 26 | 4.13 (5.50)
  Week 52: number analyzed (Participants) | 19
  Week 52 | 2.46 (4.39)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug in the parent study (20120331) through 30 days after the last dose in the extension study; actual median duration of treatment was 439 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=30)
Anaemia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Arteriovenous fistula site infection (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Endocarditis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
HIV infection (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Fluid overload (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Exsanguination (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=30)
Anaemia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 2
Catheter site haemorrhage (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 3
Seasonal allergy (Immune system disorders) | 4
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 9
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 3
Procedural vomiting (Injury, poisoning and procedural complications) | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 2
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2
Blood calcium decreased (Investigations) | 10
Blood parathyroid hormone decreased (Investigations) | 2
Blood pressure increased (Investigations) | 2
Fluid overload (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2
Venous stenosis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.